CLINICAL TRIAL: NCT01821625
Title: Study of Quadruple Therapy With Eltrombopag for Chronic Hepatitis C
Acronym: SQUELCH-C
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Interferon use for hepatitis C plummeted, eliminating the need for study drug.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 032013-020
Record Dates: First submitted 2013-03-23; First posted 2013-04-01 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Thrombocytopenia; Hepatitis C
Keywords: Thrombocytopenia; Hepatitis; Platelets; Eltrombopag; Liver Disease; Antiviral Treatment
MeSH Terms: conditions — Thrombocytopenia; Hepatitis C; Hepatitis; Liver Diseases | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thrombocytopenic (Low Platelet) Patients (Experimental): All study patients will undergo intervention in this study.
  The intervention will be a lead-in with eltrombopag and antiviral triple therapy (interferon, ribavirin and boceprevir).
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Study patients will be provided eltrombopag to raise platelet levels before anti-hepatitis C drugs are initiated, and will continue eltrombopag throughout the study.
  Other Names: Promacta

SUMMARY:
This study will provide chronic hepatitis C patients with low platelets (less than 75x10^9/L) the opportunity to undergo treatment and possible cure of their virus. The main hepatitis C drugs will be administered as standard of care, with the addition of the study drug eltrombopag.

The investigators hypothesize that providing eltrombopag to chronic hepatitis C patients with low platelets (less than 75x10^9/L) will permit the initiation and completion of antiviral triple therapy with boceprevir, ribavirin, and pegylated-interferon.

DETAILED DESCRIPTION:
SQUELCH-C is an investigator-initiated, single arm, non-blinded pilot study on the use of eltrombopag in combination with ribavirin, pegylated-interferon, and boceprevir, for patients who would not otherwise be treatment candidates because of low platelet counts (less than 75x10^9/L).

Administration of the drugs ribavirin and boceprevir will be standard of care, with one exception for interferon.

The total drug treatment period for the study patient will range from 32 - 56 weeks, depending on liver disease stage and viral response. Follow-up will take place at 12 and 24 weeks post treatment to evaluate for sustained viral response. Total study participation may require 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at least 18 years of age.
* Require a platelet count below 75 x 10^9 /L at time of screening.
* The patients must meet the eligibility criteria for all drugs involved.
* Only genotype 1 (a, b, indeterminate, or mixed).
* Confirmed history of chronic hepatitis C.
* Cirrhotic patients will be included.
* Liver imaging within 1 year to exclude hepatocellular carcinoma (HCC) is required in patients with cirrhosis.
* Patients without evidence of cirrhosis but meeting platelet criteria will also be admitted to study.
* Subjects must be able to provide informed consent, comply with drug administration instructions, and be able to complete each study visit.
* Ability to cover costs of ribavirin, interferon, and boceprevir will also be required.
* Female subjects are eligible if: Non-pregnant, non-childbearing potential, or of childbearing potential and willing to perform complete abstinence or correctly use a form of birth control during intercourse [barrier method, intrauterine device, hormonal therapy, or surgical sterilization in females or male partner]. They must also be willing to have pregnancy tests performed every 4- weeks until 6 months after completion of ribavirin.
* Male study participants must agree to use a condom and their female partner must partake in one of the contraceptive methods discussed above until 6 months after completion of ribavirin therapy.

Exclusion Criteria:

* A history of chronic infection (i.e., HIV or HBV) or a previous organ transplantation.
* A history of a platelet disorder.
* A poorly controlled underlying medical illness (i.e., diabetes, hypertension, coronary artery disease, congestive heart failure, etc.).
* Any contraindication to any study drugs as mentioned in their respective prescribing information.
* Patients with decompensated cirrhosis defined as current evidence for ascites, encephalopathy, infection or variceal bleeding. All patients should be considered Child-Pugh Class A.
* Patients with aminotransferase levels ≥ 500 IU/L will be excluded on presumption of another active liver disease.
* Patients must not be pregnant or nursing.
* The study physician maintains the right to exclude a patient for a medical condition not listed above or based off laboratory values indicating chronic disease discovered at screening.
* Patients with eye disease may be excluded from this study if the ophthalmologist does not recommend treatment.
* Subjects with known hypersensitivity reactions (such as Stevens-Johnson syndrome, toxic, epidermal necrolysis, and erythema multiforme to ribavirin) to study drugs or any component of the products.
* Subjects with autoimmune hepatitis, hemoglobinopathies (e.g., thalassemia major, sickle-cell anemia), creatinine clearance less than 50 mL/min.
* Co-administration of drugs that are highly dependent on CYP3A4/5 for clearance and CYP3A4/5 inducers (See Table 2 in boceprevir prescribing information).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M Lee, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Thrombocytopenic (Low Platelet) Patients: All study patients will undergo intervention in this study.
  The intervention will be a lead-in with eltrombopag and antiviral triple therapy (interferon, ribavirin and boceprevir).
  Eltrombopag: Study patients will be provided eltrombopag to raise platelet levels before anti-hepatitis C drugs are initiated, and will continue eltrombopag throughout the study.
Period: Overall Study
Arm/Group | Thrombocytopenic (Low Platelet) Patients
Started | 7
Completed | 1
Not Completed | 6
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 1
Not completed — Medical contraindication | 1

BASELINE CHARACTERISTICS:
Arm/Group | Thrombocytopenic (Low Platelet) Patients
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [52 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Study Patients Completing Antiviral Therapy, as Per Boceprevir Prescribing Guidelines.
Description: The length of therapy will depend on several factors:
  1. Study patient's liver disease status.
  2. Study patient's antiviral response.
  3. Study patient's tolerance to treatment.
  One patient completed therapy and experienced a sustained viral response.
  A minimum full course of treatment will be 30 weeks, with a maximum of 56 weeks of treatment.
Time Frame: Up to 56 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Thrombocytopenic (Low Platelet) Patients
Number analyzed (Participants) | 7
Participants | 1

ADVERSE EVENTS:
Time Frame: 24 months
Description: No unusual collection of adverse events.
Groups:
- Thrombocytopenic (Low Platelet) Patients: All study patients will undergo intervention in this study.
  The intervention will be a lead-in with eltrombopag and antiviral triple therapy (interferon, ribavirin and boceprevir).
  Eltrombopag: Study patients will be provided eltrombopag to raise platelet levels before anti-hepatitis C drugs are initiated, and will continue eltrombopag throughout the study.
  One subject completed the study as planned. Four subjects had to drop out of the study early for different reasons. One subject was not able to start the hepatitis C triple therapy medications due to a medical condition, two subjects discontinued due to lack of virologic response and one subject discontinued treatment due to side effects.
Arm/Group | Thrombocytopenic (Low Platelet) Patients
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thrombocytopenic (Low Platelet) Patients (N=7)
Variceal hemorrhage (Gastrointestinal disorders) | 1 (1) — Self-limited GI bleeding as can be seen in cirrhosis.
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) — prior skin ulcer on leg exacerbation
Flu like symptoms (Nervous system disorders) | 1 (1) — Flu like symptoms due to interferon therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No